CLINICAL TRIAL: NCT02142335
Title: A Phase II Trial of the Combination of Rituxan and Abraxane for the Treatment of Patients With Inoperable Stage III and IV Malignant Melanoma
Brief Title: Rituxan and Abraxane for the Treatment of Patients With Inoperable Stage III and IV Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Cancer Assocaties for Research & Excellence (Other)
Responsible Party: Principal Investigator, Edward F. McClay, M.D., Principal Investigator, California Cancer Assocaties for Research & Excellence
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29065; 20132169 (Other: WIRB)
Record Dates: First submitted 2014-03-25; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Malignant Melanoma of Skin Stage III; Metastatic Melanoma
Keywords: B-Raf, inoperable stage III melanoma, metastatic stage IV melanoma,
MeSH Terms: conditions — Melanoma | interventions — Rituximab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituxan/Abraxane (Experimental): This is a single arm study. All patients recieve treatment.
  Interventions: Drug: Rituxan

INTERVENTIONS:
Drug: Rituxan — The dose of Rituxan is 375 mg/m2¬ administered as an IV infusion during weeks 1 & 3 (days 1 & 15)Abraxane will be administered at a fixed dose of 100 mg/m2 as an IV infusion weekly for three weeks in a row followed by one week of rest
  Other Names: Abraxane

SUMMARY:
The purpose of this research study is to test an experimental combination of drugs to determine if they can cause shrinkage or even complete disappearance of your melanoma. The two drugs being tested in combination are Rituxan and Abraxane

DETAILED DESCRIPTION:
Rituxan and Abraxane are approved for the treatment of other cancers, but not for melanoma. Candidates for this study have melanoma that has spread to their lymph nodes or internal organs and that cannot be removed by a surgical procedure.

The safety of this combination of drugs will also be looked at throughout this study.

Rituxan will be administered IV at weeks 1 and 3 of each cycle. Abraxane will be administered IV weekly for 3 consecutive weeks. This is followed by 1 week of rest after which, the cycle is repeated. Following the second cycle, there will be a 4-week period of rest. Evaluation of response will occur on day 71 +/-3 days. If either disease stabilization or clear evidence of clinical response is observed two additional cycles of treatment will be administered. Lesions will be measured on the scan (CT or PET/CT), x-ray

ELIGIBILITY:
Inclusion Criteria:

* Patients must have inoperable stage III and IV melanoma.

Patients will be included in the trial based on the following criteria:

Patients previously treated with no more than 1 non-abraxane containing chemotherapy regimen or patients with the B-Raf mutation, who have received vemurafenib or the combination of Dabrafinib and trametinib (or similar compound on clinical trial) and progressed, who have documented surgically inoperable stage III or IV metastatic melanoma on pathologic examination of tissue. Previous treatment with immunotherapy is allowed. Patients who have been treated with either immunotherapy or chemotherapy must have be either 4 weeks from their last treatment or have fully recovered from all previous treatment.

Measurable or evaluable non-CNS disease required as defined:

* Uni-dimensionally measurable lesion as determined by physical exam, X-ray, CT scan, MRI, or other radiographic procedure.
* Lesion that can be seen on a radiologic test but is not uni-dimensionally measurable
* Previously irradiated lesion allowed only with documentation of progression if no other metastatic site present.

No active brain metastases Patients with previously treated brain metastases that have responded to therapy will be allowed on study assuming there is measurable disease outside of the CNS. Active therapy for the CNS disease must be completed a minimum of 3 weeks for chemotherapy and 6 weeks for radiation therapy (prior to enrollment on this study).

Prior/ Concurrent therapy

Biologic therapy No concurrent biological therapy with the exception of growth factors for anemia, neutropenia or thrombocytopenia.

Chemotherapy No greater than 1 previous non-abraxane containing chemotherapy treatment allowed

Radiotherapy At least 6 weeks since completion of radiotherapy

Patient characteristics Age and ability to give informed consent Patients must be 18 years of age or older. Patients must have the ability to give informed consent.

Performance status ECOG 0-2 Life expectancy of at least 3 months

General Medical Concerns:

* Normal organ function, except if abnormal due to tumor involvement.
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
* Subject has provided written informed consent.

Rituximab-Specific Concerns:

* ANC: > 1200/mm3
* Platelets: > 100,000/mm3
* Hemoglobin: > 9 gm/dL
* Adequate renal function as indicated by serum creatinine measurement < 1.5 x the upper limit of normal or GFR > 50 ml/min.
* Adequate liver function, as indicated by bilirubin < 3.0
* AST or ALT <2x Upper Limit of Normal unless related to primary disease.
* AST or ALT <5x Upper limit of Normal if evidence of liver metastasis.

Exclusion Criteria:

* Life expectancy less than 3 months

Untreated brain metastasis

Previous treatment with Abraxane containing regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Overall response as determined by a Percent change (%) in the sum of the diameters of target lesions. | baseline-12 weeks
  Evaluation of response (Progression Free and overall survival will be determined by measuring and recording the largest diameter of a lesion. Add these values together and record the value as the sum of the largest diameters.The percent change will be obtained according to the following formula:
  Percent change = sum of the longest diameter at 12weeks X 100 Sum of the longest diameters pre treatment

SECONDARY OUTCOMES:
Response rate as Percent change in diameter (mm) of target lesions | 2 years
  Overall response rate ( complete response + Partial response) will be determined by the disappearance of lesions or a reduction of target lesions in short axis to <10mm (CR) + at least a 30% decrease in the sum of the longest diameters of the target lesions (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. McClay, M.D., Principal Investigator — California Cancer Assocaties for Research & Excellence
Locations (1):
- California Cancer Associates For Research,cCARE, Encinitas, California, United States

REFERENCES:
- See also: California Cancer Associates For Research and Excellence, ccare clinical trials — http://pacificoncology.com/